CLINICAL TRIAL: NCT06448091
Title: Trial of Precision Medicine in Emergency Departments
Acronym: TOPMEDs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202301675; R01HG013416 (NIH)
Record Dates: First submitted 2024-05-31; First posted 2024-06-07 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Pharmacogenomic Drug Interaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Immediate panel-based pharmacogenetic genotyping (Experimental): Subjects assigned to the immediate pharmacogenetic genotyping group will be tested and have their results both entered into their electronic health record as well as provided to them within 2-4 weeks from randomization.
  Interventions: Diagnostic Test: Panel-based pharmacogenetic genotyping
- Delayed panel-based pharmacogenetic genotyping (No Intervention): Subjects assigned to delayed panel-based pharmacogenetic genotyping will not be tested until after their participation in the study has ended (6 months after enrollment).

INTERVENTIONS:
Diagnostic Test: Panel-based pharmacogenetic genotyping — After consent and randomization into the immediate PGx testing, participants' results will (10-14 days after randomization) go into their EHR and be returned via a laminated results card
  Arms: Experimental: Immediate panel-based pharmacogenetic genotyping

SUMMARY:
The objectives of this study are to (1) test the feasibility of the clinical implementation of preemptive pharmacogenetic (PGx) testing in the emergency department (ED) and (2) determine if PGx testing (with appropriate decision support) decreases ED return visits and hospitalizations. We will conduct a randomized, controlled, pragmatic clinical trial assessing both the real-world effectiveness as well as implementation outcomes using a targeted PGx testing panel in several UF Health EDs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 40 years or older presenting to a participating ED
2. Receipt of a new order/prescription for a selected PGx medication (Appendix 1), with a duration greater than 7 days, during the current ED visit or within 30 days prior.
3. Documentation of at least 2 prior ED or urgent care visits within the past 12 months

Exclusion Criteria:

1. Prior clinical pharmacogenetic test results within the EHR for genes relevant for this study (Appendix 1).
2. History of hepatic or renal transplant
3. History of severe liver disease (stage Child-Pugh C) or renal disease eGFR <15 ml/min.
4. Any medical condition that would prohibit the ability to complete the study
5. Prisoners, wards of the state, or patients being held under the Baker Act or Marchman Act
6. Life expectancy less than 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
ED recidivism | Baseline to 6 months
  The primary effectiveness outcome for the trial will be ED recidivism between participants assigned to PGx testing (intervention) compared to those assigned to delayed genotyping (usual care) within 6 months. Specifically, the rate of return visits related to their prior medical problem, identified through a matching primary diagnosis code or clinical impression abstracted from the EHR.
Rate of Clinician review of PGx results | Return of Results to 6-months
  The primary implementation outcome will be the rate at which clinicians review the PGx results. This will include both viewing of CDS alerts within the UF Health EHR or viewing individualized PGx recommendations routed from patient PGx results cards.

CONTACTS AND LOCATIONS:
Overall Officials: Julio D Duarte, Pharm.D., Ph.D., Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - UF Health Emergency Department, Gainesville, Florida
  - UF Health Jacksonville Downtown Emergency Department, Jacksonville, Florida
  - UF Health Jacksonville North Emergency Department, Jacksonville, Florida